CLINICAL TRIAL: NCT06883526
Title: A Multicenter, Open-Label, Dose-Escalation and Dose-Expansion Phase I/II Study of ZG005 in Combination With Gecacitinib in Patients With Relapsed or Refractory Lymphoma
Brief Title: Study of ZG005 in Combination With Gecacitinib in Patients With Relapsed or Refractory Lymphoma
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Suzhou Zelgen Biopharmaceuticals Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ZG005-JAK-002
Record Dates: First submitted 2025-03-13; First posted 2025-03-19 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-04

CONDITIONS: Lymphoma
MeSH Terms: conditions — Lymphoma | interventions — Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Part 1: Plan A (Experimental): ZG005（20mg/kg Q3W）+Gecacitinib（Gecacitinib is administered continuously until the end of treatment）
  Interventions: Biological: ZG005 for Injection; Drug: Gecacitinib Hydrochloride Tablets
- Part 1: Plan B (Experimental): ZG005（20mg/kg Q3W）+Gecacitinib（Gecacitinib is administered continuously from CnD1 to D14, and discontinued from CnD15 to D21）
  Interventions: Biological: ZG005 for Injection; Drug: Gecacitinib Hydrochloride Tablets

INTERVENTIONS:
Biological: ZG005 for Injection — intravenous infusion
  Other Names: ZG005
Drug: Gecacitinib Hydrochloride Tablets — Oral
  Other Names: Gecacitinib

SUMMARY:
PART 1:

1. To explore the safety of ZG005 in combination with Gecacitinib in patients with relapsed or refractory lymphoma.
2. To determine the recommended Phase II dosing regimen for relapsed or refractory lymphoma.

PART 2:

To evaluate the efficacy of ZG005 in combination with Gecacitinib in patients with relapsed or refractory lymphoma.

ELIGIBILITY:
Inclusion Criteria:

* Fully understand this study and voluntarily sign the ICF；
* Age ≥18 at ICF signing, regardless of gender；
* Histologically confirmed relapsed or refractory lymphoma.

Exclusion Criteria:

* Lymphoma with known CNS involvement；
* Severe cardiovascular/cerebrovascular diseases.
* Any other reason deeming the participant unsuitable for the study, as judged by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-05-16 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | Up to 2 years

SECONDARY OUTCOMES:
Immunogenicity | Up to 2 years
  Incidence of antidrug antibodies (ADA)

CONTACTS AND LOCATIONS:
Overall Officials: Jason Wu, Study Chair — Suzhou Zelgen Biopharmaceuticals Co.,Ltd
Locations (1):
- The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No